CLINICAL TRIAL: NCT02858388
Title: Safety and Efficacy of Sinuclean Nebules 45 (Class 1 Medical Device) in the Treatment of Pediatric Exudative Otitis Media, Randomized, Double Blind, Comparative, Parallel Study
Brief Title: Sinuclean Nebules 45 for Treatment of Pediatric Exudative Otitis Media
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galsor S.r.l. (Industry)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OME01-2014
Record Dates: First submitted 2016-06-26; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Otitis Media With Effusion
Keywords: Otitis Media with Effusion; Exudative otitis media
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SN45 (Active Comparator): Sinuclean Nebules 45
  Interventions: Device: Sinuclean Nebules 45
- Sal (Placebo Comparator): Saline solution
  Interventions: Other: Saline solution

INTERVENTIONS:
Device: Sinuclean Nebules 45 — Nebulization of solution
  Arms: SN45
Other: Saline solution — Nebulization of solution
  Arms: Sal

SUMMARY:
The goal of the study is to investigate if the active agent of Sinuclean Nebules is efficacious in the treatment of pediatric exudative otitis media, comparing with saline.

Sinuclean Nebules is a solution of cucurbitacins B,D,I,E (glycosylated triterpenes) 45 mcg, extracted from Ecballium Elaterium.

DETAILED DESCRIPTION:
Eligible pediatric subjects with diagnosis of mono or bi-lateral exudative otitis media (obtained with otorhinolaryngologic endoscopic examination, tympanogram and tonal audiometry), are randomized to treatment with Sinuclean Nebules 45 or saline.

Treatment is administered by trained caregiver with nebulizer (Rinowash Nasal Shower): one nebulization/nostril/day for two cycles of 10 consecutive days. Cycles are interrupted by a period of 7 days.

Visits 1 Baseline T0: confirmation of eligibility, randomization, training of caregiver, dispensation of blinded therapy for two cycles, delivery of the clinical diary.

Visit 2 after 10 days of therapy + 7 days of interval: phone call to check for adverse events, therapy adherence, concomitant diseases and treatments, and to prescribe second cycle of therapy.

Visit 3 End of Study: assessment of the exudative otitis media with otorhinolaryngologic endoscopic examination, tympanogram tonal audiometry, verification of the subject's clinical diary.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of mono or bi-lateral exudative otitis media, performed the day of recruitment or in the week before, with endotympanic effusion present for at least 3 months, and hearing loss.
* The diagnostic criteria is type B tympanogram for at least one of the two ears.
* The criteria is integrated by a) tonal audiometry to demonstrate bilateral or monolateral deficit (loss of more than 20dB averaged to 0.5-1.2 and 4Khz in the best ear with pure tone audiometry); for 1-3 yo subjects the audiometry is behavioural b) otorhinolaryngologic examination in endoscopy for the otologic, rhino-sinusal and pharyngeal districts.

Exclusion Criteria:

1. Outcomes of adenotonsillectomy
2. Velo-palatal insufficiencies, cleft lip and cleft palate.
3. Hearing loss of perceptual, and mixed type.
4. Clinical conditions (systemic diseases or other) that may interfere with the evaluation of safety and clinical effectiveness of the product under investigation, for example: diabetes mellitus, heart disease, chronic renal failure, active systemic infections)
5. Assumption, during the study of drugs that may interfere with the assessment of the product object of clinical investigation.
6. Possibility of needing treatment during the study with drugs that are not allowed, for example: antibiotics in long-term prophylaxis, immunosuppressants, corticosteroids.
7. Regular intake of steroids in the four weeks preceding the date of the admission visit.
8. Viral or allergic rhinitis, with active effusion.
9. Down Syndrome
10. Diagnosis of immotile cilia syndrome
11. Condition of immune deficiency disease or otherwise.
12. Cystic Fibrosis.
13. Dental malocclusion
14. Other diseases of other organ systems, which, in the opinion of the investigator, may interfere with the purpose or the study procedures.
15. Not vaccinated subjects, with no clinical history of varicella who have been in contact, in the 4 weeks before the admission visit, with people who may be suffering from chicken pox or Zoster.
16. Psychic condition incompatible with participation in the research.
17. History of intolerance or allergy to the components of Sinuclean Nebules.
18. Medical and surgical intervention that may prejudice the complete execution of the trial, in the 4 weeks preceding the signing of informed consent.
19. Imminence of a medical-surgical procedure that can jeopardize the completion of the trial.
20. Participation in the course to other clinical investigations, or terminated within 30 days of the start of this trial.
21. Previous randomization in the study
22. Be first- or second-grade relative of a member of the Site study staff.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Resolution of tympanic effusion | At Day 28 after start of treatment
  The resolution of the tympanic effusion will be assessed with tympanogram (% of subjects with type A tympanogram).

SECONDARY OUTCOMES:
Complete auditory recovery | At Day 28 after start of treatment
  The auditory recovery will be measured with tonal audiometry, % of subjects recovering normal values (threshold by air between 0 and 25 dB).

CONTACTS AND LOCATIONS:
Overall Officials: Attilio Varricchio, MD, Principal Investigator — San Gennaro Hospital, Naples, Italy
Locations (1):
- San Gennaro Hospital, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zielhuis GA, Straatman H, Rach GH, van den Broek P. Analysis and presentation of data on the natural course of otitis media with effusion in children. Int J Epidemiol. 1990 Dec;19(4):1037-44. doi: 10.1093/ije/19.4.1037. PMID 2083987